CLINICAL TRIAL: NCT03365752
Title: A Comparison Study to Facilitate Earlier Discharge: Spinal Versus General Anesthesia for Outpatient Knee Surgeries, a Randomized Controlled Study
Brief Title: Chloroprocaine Spinal for Outpatient Knee Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted due to COVID-19 pandemic and terminated early per request of principal investigator as Chloroprocaine use in spinal procedures has become incorporated as standard of care at HSS.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-1547
Record Dates: First submitted 2017-11-27; First posted 2017-12-07 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Knee Arthroscopy
MeSH Terms: interventions — chloroprocaine; Mepivacaine; Anesthetics, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Chloroprocaine (Experimental)
  Interventions: Drug: Chloroprocaine
- Mepivacaine (Active Comparator)
  Interventions: Drug: Mepivacaine
- General Anesthesia (Active Comparator)
  Interventions: Drug: General Anesthetics

INTERVENTIONS:
Drug: Chloroprocaine — A spinal anesthetic with 2% chloroprocaine (2cc or 40 mg) will be performed
  Arms: Chloroprocaine
Drug: Mepivacaine — A spinal anesthetic with 1.5% Mepivacaine (3cc or 45 mg) will be performed
  Arms: Mepivacaine
Drug: General Anesthetics — General anesthetics will be administered intravenously
  Arms: General Anesthesia

SUMMARY:
Outpatient knee surgeries with duration of less than one hour pose a challenge to the use of spinal anesthesia given that traditional agents remain in effect for 2-3 hours, thus creating a mismatch between length of surgery and anesthetic resolution. The investigators hypothesize that the use of chloroprocaine can combine the benefits of a short spinal anesthetic while avoiding the side effects of a general anesthetic, thus promoting earlier discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a knee arthroscopy that is anticipated to be less than one hour
* Age 18 to 80 years
* Ability to follow study protocol
* English speaking

Exclusion Criteria:

* Hepatic or renal insufficiency
* Younger than 18 years old and older than 80
* Allergy or intolerance to one of the study medications
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)
* Patients unable to undergo a spinal anesthetic or Laryngeal Mask Airway (LMA)/GA or patient refusal to spinal anesthesia or LMA/GA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-24 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kim, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chloroprocaine | Mepivacaine | General Anesthesia
Started | 13 | 13 | 13
Completed | 13 | 13 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine | Mepivacaine | General Anesthesia | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.26 (15.87) | 51.90 (12.34) | 50.65 (13.39) | 50.6 (13.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 14
  Male | 9 | 8 | 8 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 12 | 13 | 13 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 3 | 5
  White | 10 | 13 | 7 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.35 (4.79) | 27.96 (6.35) | 28.65 (4.82) | 27.99 (5.25)
ASA Physical Status Classification [Count of Participants; unit: Participants]
  ASA I - A normal healthy patient | 4 | 1 | 4 | 9
  ASA II - A patient with mild systemic disease | 9 | 12 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Readiness for Discharge
Description: Defined as duration from arrival in the post-anesthesia care unit (PACU0 to the time patient meets the discharge criteria from the post anesthesia discharge scoring system (PADSS) for home readiness after ambulatory surgery
Time Frame: Determine within 24 hours after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Mepivacaine | General Anesthesia
Number analyzed (Participants) | 13 | 13 | 13
minutes | 141.85 (39.17) | 174.31 (38.74) | 170.69 (67.9)

ADVERSE EVENTS:
Time Frame: Safety surveillance and reporting starts as soon as the subject undergoes surgery and receives treatment and lasts until the subject concludes their participation in the study or the subject/investigator withdraws the subject from the study. Up to 7 days following surgery.
Arm/Group | Chloroprocaine | Mepivacaine | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
This project was terminated early, as enrollment was negatively impacted to due to the COVID-19 pandemic and because clinical practice has shifted to include the use of chloroprocaine in spinal procedures as standard of care at the Hospital for Special Surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT03365752/Prot_SAP_000.pdf